CLINICAL TRIAL: NCT00999141
Title: A Randomized, Controlled Phase 3 Study to Evaluate Safety and Efficacy of Fibrin Sealant (FS) VH S/D 4 S-apr (ARTISS) to Adhere Tissues and Improve Wound Healing in Subjects Undergoing Rhytidectomy (Facelift)
Brief Title: Efficacy and Safety of FS VH S/D 4 S-apr for Flap Adherence in Rhytidectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 550901
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Face-lift; Facial Rhytidectomy
MeSH Terms: interventions — Low Density Lipoprotein Receptor-Related Protein-1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FS VH S/D 4 s-apr (Experimental): One side of face will be treated with the investigational product (FS VH S/D 4 s-apr) as an adjuvant to the standard of care. Please note: Each subject will participate in both arms (investigational product and standard of care) simultaneously, and will serve as his/her own control.
  Interventions: Biological: FS VH S/D 4 s-apr
- Standard of Care (SoC) (No Intervention): Other side of face will receive standard of care. Please note: Each subject will participate in both arms (investigational product and standard of care) simultaneously, and will serve as his/her own control.

INTERVENTIONS:
Biological: FS VH S/D 4 s-apr — FS VH S/D 4 s-apr will be applied (using spray device provided by Sponsor) to the subcutaneous plane (intraoperative, topical administration) in both the neck and the face area.
  Other Names: ARTISS
  Arms: FS VH S/D 4 s-apr

SUMMARY:
The purpose of the study is to compare the safety and efficacy of FS VH S/D 4 s-apr versus standard of care in adhering tissue and improving wound healing in subjects undergoing facelift.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject is 18 to 75 years of age at the time of screening
* Subject is planned for facial rhytidectomy
* Subject has read, understood and signed the written informed consent
* Subject is healthy, as determined by the investigator using standard pre-operative assessments to include laboratory tests and electrocardiograms
* Subject is of childbearing potential, presents with a negative serum pregnancy test, and agrees to employ adequate birth control measures for the duration of the study
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Subject is indicated for an abbreviated or modified face-lift procedure such as deep plane procedures, minimal undermining procedures, thread lifts, and minimal access cranial suspension
* Subject is indicated for concurrent facial surgeries during the operation (eg forehead plasty,blepharoplasty, rhinoplasty, buccal fat removal, any filler injections including fat injections, lip augmentation, skin resurfacing procedures etc.)
* Subject is indicated for additional procedures to the body during the same operation (eg liposuction, mastoplasty etc.)
* Subject has undergone a prior rhytidectomy surgery
* Subject is an active smoker, as assessed by the investigator
* Subject has a known (documented) bleeding or coagulation disorder
* Subject is being treated with anti-coagulants or with Aspirin (that was not discontinued 7 days prior to surgery)
* Subject has a vascular disorder, cardiovascular disease, and/or uncontrolled hypertension
* Subject has diabetes mellitus with glycosylated hemoglobin (HbA1c) > 7
* Subject is receiving active treatment for a malignancy
* Subject has a connective tissue disorder
* Subject has an active or chronic skin disorder
* Subject has history of Bell's palsy
* Subject has a documented history of pathologically or pharmacologically induced immune deficiency
* Subject has received chronic treatment with immunosuppressive drugs, systemic corticosteroids, or other chronic treatments within 30 days prior to the surgery
* Subject has a known sensitivity to components of FS VH S/D 4 s-apr
* Subject has a known psychiatric disorder (eg, obsessive compulsive disorder, anxiety, eating disorders, etc.)
* Subject has documented healing complications following previous surgeries (eg, hypertrophic scarring)
* Subject is pregnant or lactating at the time of enrollment
* Subject has participated in another clinical study involving an investigational product/device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an investigational product/device during the course of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Z Abrams, MD, Study Director — Baxter Healthcare Corporation
Locations (6):
- United States (6):
  - Beverly Hills, California
  - Atlanta, Georgia
  - Evans, Georgia
  - Hewlett, New York
  - Chattanooga, Tennessee
  - Dallas, Texas

REFERENCES:
- [Derived] Hester TR Jr, Shire JR, Nguyen DB, Gerut ZE, Chen AH, Diamond J, Desmond JC, Silvati-Fidell L, Abrams SZ, Rohrich RJ. Randomized, controlled, phase 3 study to evaluate the safety and efficacy of fibrin sealant VH S/D 4 s-apr (Artiss) to improve tissue adherence in subjects undergoing rhytidectomy. Aesthet Surg J. 2013 May;33(4):487-96. doi: 10.1177/1090820X13479969. Epub 2013 Apr 5. PMID 23563904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 7 clinical sites in the United States, beginning September 2009 and completing in December 2009
Pre-assignment Details: 79 participants were enrolled and screened. 2 were screen failures and 2 requested withdrawal. Therefore, 75 of the 79 enrolled were randomized.
Groups:
- Facelift Participants: One side of face will be treated with the investigational product (FS VH S/D 4 s-apr) as an adjuvant to the standard of care (SoC), and the other side of the face will receive SoC alone. Please note: Each subject will participate in both arms (investigational product and SoC) simultaneously, and will serve as his/her own control.
Period: Overall Study
Arm/Group | Facelift Participants
Started | 75 (Randomized and treated)
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Facelift Participants
Number analyzed (Participants) | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Total Volume of Drainage on Each Side of the Face
Description: Total drainage volume collected from each side of the face. One side of face is treated with FS VH S/D 4 s-apr (FS); the other side is treated using standard of care (SoC).
Time Frame: 24 hours (± 4h) after surgery
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Median (Full Range); unit: mL
Arm/Group | Standard of Care (SoC) | FS VH S/D 4 S-apr
Number analyzed (Participants) | 75 | 75
mL | 20.0 [0 to 50] | 8.0 [0 to 39]
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FS VH S/D 4 S-apr; Test type: Superiority or Other; p < 0.0001, two-sided paired t-test; alpha = 5%

2. Secondary Outcome: Participants' First Occurrence of Hematoma or Seroma by Study Day
Description: Investigators assessed each side of the face for the presence of hematomas and/or seromas
Time Frame: Day 0 (day of surgery) through postoperative day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | FS VH S/D 4 S-apr Side - Hematoma | FS VH S/D 4 S-apr Side - Seroma | Standard of Care (SoC) Side - Hematoma | Standard of Care (SoC) Side - Seroma
Number analyzed (Participants) | 75 | 75 | 75 | 75
participants
  Day 0 | 0 | 0 | 1 | 0
  Day 1 | 1 | 2 | 0 | 1
  Day 2 | 0 | 0 | 0 | 0
  Day 3 | 0 | 1 | 2 | 2
  Day 4 | 0 | 0 | 0 | 0
  Day 5 | 0 | 0 | 0 | 0
  Day 6 | 0 | 0 | 0 | 0
  Day 7 | 0 | 1 | 1 | 1
  Day 8 | 0 | 0 | 0 | 0
  Day 9 | 0 | 0 | 0 | 0
  Day 10 | 0 | 1 | 0 | 0
  Day 11 | 0 | 0 | 0 | 0
  Day 12 | 0 | 0 | 0 | 0
  Day 13 | 0 | 0 | 0 | 0
  Day 14 | 0 | 1 | 0 | 0

3. Secondary Outcome: Participants With Hematoma/Seroma by Study Day
Description: Investigators assessed each side of the face for the presence of hematoma and/or seroma
Time Frame: Day 0 (day of surgery) through postoperative day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Groups:
- FS VH S/D 4 S-apr: Participants With Hematoma/Seroma on FS VH S/D 4 s-apr Side
- Standard of Care (SoC): Participants With Hematoma/Seroma on SoC Side
Arm/Group | FS VH S/D 4 S-apr | Standard of Care (SoC)
Number analyzed (Participants) | 75 | 75
participants
  Day 0 | 0 | 1
  Day 1 | 3 | 1
  Day 2 | 2 | 1
  Day 3 | 2 | 4
  Day 4 | 1 | 4
  Day 5 | 0 | 3
  Day 6 | 0 | 0
  Day 7 | 1 | 2
  Day 8 | 1 | 2
  Day 9 | 1 | 2
  Day 10 | 2 | 2
  Day 11 | 0 | 1
  Day 12 | 0 | 1
  Day 13 | 0 | 1
  Day 14 | 1 | 1

4. Secondary Outcome: Number of Participants With Hematoma/Seroma Anytime During the Study
Time Frame: Day 0 (day of surgery) through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Participants With Hematoma/Seroma on FS VH S/D 4 S-apr Side | Participants With Hematoma/Seroma on SoC Side | Participants With Hematoma/Seroma on Both Sides | Participants With No Hematoma/Seroma on Either Side
Number analyzed (Participants) | 75 | 75 | 75 | 75
participants | 2 | 5 | 3 | 65
Statistical Analysis 1: Comparison: Participants With Hematoma/Seroma on FS VH S/D 4 S-apr Side vs Participants With Hematoma/Seroma on SoC Side; Test type: Superiority or Other; p = 0.257, McNemar; alpha = 5%; Difference in Proportions = 0.040, 95% CI [-0.039 to 0.125] — Difference in Proportions = (SoC) - (FS VH S/D 4 s-apr)

5. Secondary Outcome: Investigators' Visual Comparisons of Edema Between the 2 Sides of Face at Day 1
Description: Investigators' assessed which side of the face (FS VH S/D 4 s-apr or Standard SoC) had less edema
Time Frame: Through postoperative Day 1
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Participants With Less Edema on FS VH S/D 4 S-apr Side | Participants With Less Edema on SoC Side | Participants With No Difference in Edema
Number analyzed (Participants) | 75 | 75 | 75
participants | 40 | 12 | 23
Statistical Analysis 1: Comparison: Participants With Less Edema on FS VH S/D 4 S-apr Side vs Participants With Less Edema on SoC Side; Test type: Superiority or Other; p < 0.001, McNemar; alpha = 5%; Difference in proportions = -0.373, 95% CI [-0.524 to -0.193] — Difference in proportions = SoC - FS VH S/D 4 s-apr

6. Secondary Outcome: Investigators' Visual Comparisons of Edema Between the 2 Sides of Face at Day 3
Description: Investigators' assessed which side of the face (FS VH S/D 4 s-apr or Standard SoC) had less edema
Time Frame: Through postoperative Day 3
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Participants With Less Edema on FS VH S/D 4 S-apr Side | Participants With Less Edema on SoC Side | Participants With No Difference in Edema
Number analyzed (Participants) | 75 | 75 | 75
participants | 41 | 12 | 22
Statistical Analysis 1: Comparison: Participants With Less Edema on FS VH S/D 4 S-apr Side vs Participants With Less Edema on SoC Side; Test type: Superiority or Other; p < 0.001, McNemar; Difference in proportions = -0.387, 95% CI [-0.538 to -0.205] — Difference in Proportions = SoC - FS VH S/D 4 s-apr

7. Secondary Outcome: Investigators' Visual Comparisons of Edema Between the 2 Sides of Face at Day 7
Description: Investigators' assessed which side of the face (FS VH S/D 4 s-apr or Standard SoC) had less edema
Time Frame: Through postoperative Day 7
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Participants With Less Edema on FS VH S/D 4 S-apr Side | Participants With Less Edema on SoC Side | Participants With No Difference in Edema
Number analyzed (Participants) | 73 | 73 | 73
participants | 41 | 15 | 17
Statistical Analysis 1: Comparison: Participants With Less Edema on FS VH S/D 4 S-apr Side vs Participants With Less Edema on SoC Side; Test type: Superiority or Other; p = 0.001, McNemar; alpha = 5%; Difference in proportions = -0.356, 95% CI [-0.521 to -0.161] — Difference in proportions = SoC - FS VH S/D 4 s-apr

8. Secondary Outcome: Investigators' Visual Comparisons of Edema Between the 2 Sides of Face at Day 14
Description: Investigators' assessed which side of the face (FS VH S/D 4 s-apr or Standard SoC) had less edema
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Participants With Less Edema on FS VH S/D 4 S-apr Side | Participants With Less Edema on SoC Side | Participants With No Difference in Edema
Number analyzed (Participants) | 74 | 74 | 74
participants | 27 | 13 | 34
Statistical Analysis 1: Comparison: Participants With Less Edema on FS VH S/D 4 S-apr Side vs Participants With Less Edema on SoC Side; Test type: Superiority or Other; p = 0.027, McNemar; alpha = 5%; Difference in proportions = -0.189, 95% CI [-0.342 to -0.023] — Difference in proportions = SoC - FS VH S/D 4 s-apr

9. Secondary Outcome: Change From Baseline (Day 0, Preoperative) in Skin Sensitivity on Postoperative Days 3, 7, 14
Description: Skin sensitivity was measured using Semmes-Weinstein Monofilament set to detect neurological damage. Filament sizes are noted by handle numbers of measuring tools ([handle number = log10(10*force in milligrams applied to skin)], range = 1.65 to 6.65). Detection of filament with smaller handle number = greater skin sensitivity. Smaller change in filament size detection from pre-op to post-op = less impact to recovery of sensation. Smallest filament felt for each side of face was noted. Change in skin sensitivity computed as (Handle Number Postop Day 3, 7, or 14) - (Handle Number Preop Day 0).
Time Frame: Day 0 (preoperative) through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Mean (95% Confidence Interval); unit: Handle number(s)
Arm/Group | FS VH S/D 4 S-apr | Standard of Care (SoC)
Number analyzed (Participants) | 75 | 75
Handle number(s)
  Day 3 | 0.54 (0.85) [0.34 to 0.73] | 0.60 (0.94) [0.39 to 0.82]
  Day 7 | 0.44 (0.94) [0.22 to 0.65] | 0.51 (1.02) [0.27 to 0.74]
  Day 14 | 0.24 (0.82) [0.05 to 0.42] | 0.32 (0.96) [0.10 to 0.54]

10. Secondary Outcome: Participants' Assessment of Side of Face Preference (SoC and FS VH S/D 4) on Postoperative Days 1, 3, 7, 14
Description: Participants responded to the following question during the side of face preference assessment:
  "Which side of the face do you prefer? Left side, right side, or no preference?"
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Participants Preferring FS VH S/D 4 S-apr | Participants Preferring SoC | Participants With No Preference
Number analyzed (Participants) | 75 | 75 | 75
participants
  Day 1 (n= 75) | 47 | 16 | 12
  Day 3 (n= 75) | 40 | 23 | 12
  Day 7 (n= 75) | 44 | 18 | 13
  Day 14 (n= 74) | 42 | 15 | 17

11. Secondary Outcome: Proportion of Participants Preferring Either FS VH S/D 4 S-apr or SoC Side of Face - Day 1
Description: as for outcome 10
Time Frame: Through postoperative Day 1
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: Proportion of Participants
Arm/Group | Proportion of Participants Preferring FS VH S/D 4 S-apr Side | Proportion of Participants Preferring SoC Side
Number analyzed (Participants) | 75 | 75
Proportion of Participants | 0.63 | 0.21
Statistical Analysis 1: Comparison: Proportion of Participants Preferring FS VH S/D 4 S-apr Side vs Proportion of Participants Preferring SoC Side; Test type: Superiority or Other; Difference in Proportions = -0.413, 95% CI [-0.577 to -0.213] — Difference in Proportions = (SoC) - (FS VH S/D 4 s-apr)

12. Secondary Outcome: Proportion of Participants Preferring Either FS VH S/D 4 S-apr or SoC Side of Face - Day 3
Description: as for outcome 10
Time Frame: Through postoperative Day 3
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: Proportion of Participants
Arm/Group | Proportion of Participants Preferring FS VH S/D 4 S-apr Side | Proportion of Participants Preferring SoC Side
Number analyzed (Participants) | 75 | 75
Proportion of Participants | 0.53 | 0.31
Statistical Analysis 1: Comparison: Proportion of Participants Preferring FS VH S/D 4 S-apr Side vs Proportion of Participants Preferring SoC Side; Test type: Superiority or Other; Difference in Proportions = -0.227, 95% CI [-0.413 to -0.020] — Difference in Proportions = (SoC) - (FS VH S/D 4 s-apr)

13. Secondary Outcome: Proportion of Participants Preferring Either FS VH S/D 4 S-apr or SoC Side of Face - Day 7
Description: as for outcome 10
Time Frame: Through postoperative Day 7
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: Proportion of Participants
Arm/Group | Proportion of Participants Preferring FS VH S/D 4 S-apr Side | Proportion of Participants Preferring SoC Side
Number analyzed (Participants) | 75 | 75
Proportion of Participants | 0.59 | 0.24
Statistical Analysis 1: Comparison: Proportion of Participants Preferring FS VH S/D 4 S-apr Side vs Proportion of Participants Preferring SoC Side; Test type: Superiority or Other; Difference in Proportions = -0.347, 95% CI [-0.518 to -0.145] — Difference in Proportions = (SoC) - (FS VH S/D 4 s-apr)

14. Secondary Outcome: Proportion of Participants Preferring Either FS VH S/D 4 S-apr or SoC Side of Face - Day 14
Description: as for outcome 10
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: Proportion of Participants
Arm/Group | Proportion of Participants Preferring FS VH S/D 4 S-apr Side | Proportion of Participants Preferring SoC Side
Number analyzed (Participants) | 74 | 74
Proportion of Participants | 0.57 | 0.20
Statistical Analysis 1: Comparison: Proportion of Participants Preferring FS VH S/D 4 S-apr Side vs Proportion of Participants Preferring SoC Side; Test type: Superiority or Other; Difference in Proportions = -0.365, 95% CI [-0.528 to -0.171] — Difference in Proportions = (SoC) - (FS VH S/D 4 s-apr)

15. Secondary Outcome: Reasons for Participants' Preferences for Side of Face
Description: Participants responded to the following questions during the side of face preference assessment:
  1. "Which side of the face do you prefer? Left side, right side, or no preference?"
  2. If "right" or "left" is chosen, participants were asked "Please mark ALL reasons for choosing this side"
     1. Better skin sensation
     2. Less numbness
     3. Looks better
     4. Less bruising
     5. Less swelling
     6. Less pain
     7. Less itching
     8. Less tingling
     9. Less feeling of "pins and needles"
     10. Other ________________ (Free Text)
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: Participants
Arm/Group | FS VH S/D 4 S-apr Side - Day 1 | SoC Side - Day 1 | FS VH S/D 4 S-apr Side - Day 3 | SoC Side - Day 3 | FS VH S/D 4 S-apr Side - Day 7 | SoC Side - Day 7 | FS VH S/D 4 S-apr Side - Day 14 | SoC Side - Day 14
Number analyzed (Participants) | 47 | 16 | 40 | 23 | 44 | 18 | 42 | 15
Participants
  Better Skin Sensation | 19 | 5 | 15 | 4 | 19 | 7 | 26 | 6
  Less Bruising | 21 | 8 | 21 | 14 | 30 | 9 | 29 | 5
  Less Feeling of Pins and Needles | 4 | 1 | 7 | 1 | 8 | 1 | 11 | 1
  Less Itching | 2 | 2 | 7 | 3 | 9 | 1 | 11 | 0
  Less Numbness | 16 | 6 | 24 | 9 | 24 | 7 | 28 | 11
  Less Pain | 23 | 7 | 22 | 8 | 26 | 5 | 25 | 4
  Less Swelling | 37 | 14 | 30 | 16 | 33 | 14 | 36 | 12
  Less Tingling | 2 | 1 | 6 | 3 | 9 | 2 | 16 | 1
  Looks Better | 35 | 13 | 32 | 19 | 37 | 13 | 35 | 12
  Other | 3 | 0 | 3 | 1 | 3 | 0 | 2 | 1

16. Other Pre Specified Outcome: Participants' Assessment of Difference in Numbness Between Two Sides of Face
Description: During each postoperative visit (Day 1, 3, 7, and 14), participants were asked:
  How would you rate your numbness on each side of your face on a scale of 0-10, with 10 being the worst numbness possible?
  Difference in scores on a scale = (SoC score) - (FS VH S/D 4 s-apr score)
  The planned and approved Statistical Analysis Plan (SAP) called for a pre-aggregation of the data whereby differences between the two sides of the face were computed first within participants to retain the inherent correlation (pairings) in the measures. Summary statistics and statistical tests were then computed on the differences between the two sides of the face using paired sample tests.
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Facelift Participants
Number analyzed (Participants) | 75
Scores on a scale
  Postoperative Day 1 | 0.3 (2.0)
  Postoperative Day 3 | 0.4 (1.7)
  Postoperative Day 7 | 0.3 (1.4)
  Postoperative Day 14 | 0.5 (1.4)

17. Other Pre Specified Outcome: Investigator Preference for Side of Face
Description: Investigator reported outcomes data was collected for overall preference for 1 side of face
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Strongly Prefer FS VH S/D 4 S-apr Side | Somewhat Prefer FS VH S/D 4 S-apr Side | No Preference | Somewhat Prefer SoC Side | Strongly Prefer SoC Side
Number analyzed (Participants) | 75 | 75 | 75 | 75 | 75
participants
  Postoperative Day 1 | 8 | 33 | 21 | 13 | 0
  Postoperative Day 3 | 7 | 37 | 18 | 10 | 3
  Postoperative Day 7 | 16 | 31 | 16 | 11 | 1
  Postoperative Day 14 | 16 | 21 | 25 | 12 | 1

18. Other Pre Specified Outcome: Investigators' Satisfaction With Quality of Flap Adherence
Description: During postoperative visits investigators recorded their satisfaction with the quality of flap adherence for each side of the face (FS VH S/D 4 s-apr (FS) or Standard of Care (SoC) sides of face)
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Not at All Satisfied | A Little Satisfied | Somewhat Satisfied | Moderately Satisfied | Very Satisfied
Number analyzed (Participants) | 75 | 75 | 75 | 75 | 75
participants
  Satisfaction with flap adherence FS Side- Day 1 | 1 | 0 | 8 | 19 | 47
  Satisfaction with flap adherence FS Side- Day 3 | 0 | 1 | 6 | 18 | 50
  Satisfaction with flap adherence FS Side- Day 7 | 0 | 0 | 1 | 14 | 60
  Satisfaction with flap adherence FS Side- Day 14 | 0 | 0 | 1 | 12 | 62
  Satisfaction with flap adherence SoC Side- Day 1 | 0 | 7 | 13 | 26 | 29
  Satisfaction with flap adherence SoC Side- Day 3 | 0 | 1 | 23 | 13 | 38
  Satisfaction with flap adherence SoC Side- Day 7 | 0 | 0 | 11 | 25 | 39
  Satisfaction with flap adherence SoC Side- Day 14 | 0 | 0 | 5 | 21 | 49

19. Other Pre Specified Outcome: Investigators' Satisfaction With Rate of Healing
Description: During postoperative visits investigators recorded their satisfaction with the rate of healing of each side of the face (FS VH S/D 4 s-apr (FS) or Standard of Care (SoC) sides of face)
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Not at All Satisfied | A Little Satisfied | Somewhat Satisfied | Moderately Satisfied | Very Satisfied
Number analyzed (Participants) | 75 | 75 | 75 | 75 | 75
participants
  Satisfaction with Rate of Healing FS Side- Day 1 | 1 | 0 | 10 | 28 | 36
  Satisfaction with Rate of Healing FS Side- Day 3 | 0 | 0 | 7 | 19 | 49
  Satisfaction with Rate of Healing FS Side- Day 7 | 0 | 0 | 1 | 14 | 60
  Satisfaction with Rate of Healing FS Side- Day 14 | 0 | 0 | 2 | 11 | 62
  Satisfaction with Rate of Healing SoC Side- Day 1 | 0 | 6 | 14 | 21 | 34
  Satisfaction with Rate of Healing SoC Side- Day 3 | 0 | 1 | 17 | 17 | 40
  Satisfaction with Rate of Healing SoC Side- Day 7 | 0 | 0 | 11 | 24 | 40
  Satisfaction with Rate of Healing SoC Side- Day 14 | 0 | 0 | 6 | 20 | 49

20. Other Pre Specified Outcome: Investigators' Satisfaction With Treatment
Description: During postoperative visits investigators recorded their satisfaction with treatment on each side of the face (FS VH S/D 4 s-apr (FS) or Standard of Care (SoC) sides of face)
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Not at All Satisfied | A Little Satisfied | Somewhat Satisfied | Moderately Satisfied | Very Satisfied
Number analyzed (Participants) | 75 | 75 | 75 | 75 | 75
participants
  Satisfaction with Treatment on FS Side- Day 1 | 1 | 0 | 7 | 19 | 48
  Satisfaction with Treatment on FS Side- Day 3 | 0 | 1 | 5 | 13 | 56
  Satisfaction with Treatment on FS Side- Day 7 | 0 | 0 | 2 | 12 | 61
  Satisfaction with Treatment on FS Side- Day 14 | 0 | 0 | 2 | 10 | 63
  Satisfaction with Treatment on SoC Side- Day 1 | 0 | 6 | 15 | 17 | 37
  Satisfaction with Treatment on SoC Side- Day 3 | 0 | 2 | 14 | 16 | 43
  Satisfaction with Treatment on SoC Side- Day 7 | 0 | 0 | 11 | 19 | 45
  Satisfaction with Treatment on SoC Side- Day 14 | 0 | 0 | 5 | 19 | 51

21. Other Pre Specified Outcome: Investigators' Confidence in Decreased Postsurgical Complications With the Use of FS VH S/D 4 S-apr
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Number; unit: participants
Arm/Group | Not Confident | Not Very Confident | Neutral | Somewhat Confident | Confident
Number analyzed (Participants) | 75 | 75 | 75 | 75 | 75
participants
  Day 1 | 0 | 0 | 8 | 20 | 47
  Day 3 | 0 | 0 | 6 | 26 | 43
  Day 7 | 0 | 0 | 5 | 20 | 50
  Day 14 | 0 | 0 | 8 | 14 | 53

22. Other Pre Specified Outcome: Total Aspiration Volumes From Hematomas and Seromas
Time Frame: Through postoperative Day 14
Population: Full Analysis Data Set = All randomized and treated participants
Measure: Median (Full Range); unit: mL
Arm/Group | FS VH S/D 4 S-apr Side - Hematoma | SoC Side - Hematoma | FS VH S/D 4 S-apr Side - Seroma | SoC Side - Seroma
Number analyzed (Participants) | 1 | 4 | 3 | 3
mL | NA [1.0 to 1.0] — The median is the central value of a series of numbers. This arm has a single data point, i.e. no series of numbers from which to determine a central value. | 4.1 [2.5 to 8.0] | 4.7 [3.0 to 12.5] | 7.0 [4.7 to 16.5]

23. Primary Outcome: Number of AEs Related to the Investigational Product (FS VH S/D 4 S-apr)
Time Frame: Day 0 (day of surgery) through postoperative Day 14
Population: Safety Analysis Set
Measure: Number; unit: Events
Arm/Group | Related Non-Facial Adverse Events | Related Facial Adverse Events
Number analyzed (Participants) | 75 | 75
Events
  Serious Adverse Events- Mild | 0 | 0
  Serious Adverse Events- Moderate | 0 | 1
  Serious Adverse Events- Severe | 0 | 0
  non-Serious Adverse Events- Mild | 0 | 2
  non-Serious Adverse Events- Moderate | 0 | 0
  non-Serious Adverse Events- Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 (day of surgery) through postoperative Day 14
Groups:
- Localized to SoC Side of Face: AE was localized to the side of the face which was treated with standard of care (SoC).
- Localized to FS VH S/D 4 S-apr Side of Face: AE was localized to the side of the face which was treated with FS VH S/D 4 s-apr
- Non-localized AEs: AE affected a site other than either side of the face (ie, non-localized AE)
Arm/Group | Localized to SoC Side of Face | Localized to FS VH S/D 4 S-apr Side of Face | Non-localized AEs
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/75 | 1/75
Other Adverse Events (participants affected / at risk) | 8/75 | 5/75 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Localized to SoC Side of Face (N=75) | Localized to FS VH S/D 4 S-apr Side of Face (N=75) | Non-localized AEs (N=75)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Localized to SoC Side of Face (N=75) | Localized to FS VH S/D 4 S-apr Side of Face (N=75) | Non-localized AEs (N=75)
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 4 (4) | 4 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of the individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥90 days prior to submission or communication. Baxter may request an additional delay of ≤60 days (e.g., for intellectual property protection)